CLINICAL TRIAL: NCT02451514
Title: A Phase 2, Open-label, Controlled, Multi-center Extension Study to Evaluate 4-year Antibody Persistence and Booster Response Following MenABCWY Vaccination in Healthy Adolescents and Young Adults Who Previously Participated in Studies V102_02 (NCT01210885) and V102_02E1 (NCT01367158)
Brief Title: A Study to Evaluate 4-year Antibody Persistence and Booster Response Following MenABCWY Vaccination in Healthy Adolescents and Young Adults Who Previously Participated in Studies V102_02 (NCT01210885) and V102_02E1 (NCT01367158)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205213; 2016-004420-29 (EudraCT Number); V102_02E2 (Other: Novartis)
Record Dates: First submitted 2015-05-04; First posted 2015-05-22 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Meningococcal Disease; Infections, Meningococcal
Keywords: Antibody persistence; Young Adults; Healthy Adolescents; MenABCWY vaccine; Booster response; MenABCWY+OMV
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MenABCWY+OMV Group (Experimental): Subjects who received 2 doses of MenABCWY+OMV vaccine in the parent study V102_02 (NCT01210885) and received no subsequent meningococcal vaccines, received a booster dose of MenABCWY+OMV vaccine in the current study at Day 1.
  Interventions: Biological: MenABCWY+OMV vaccine
- MenACWY Group (Experimental): Subjects who received MenACWY vaccine in the parent study V102_02 (NCT01210885) and received no subsequent meningococcal vaccines, received 2 doses of MenABCWY+OMV vaccine, one month apart (Day 1 and Day 31), in the current study.
  Interventions: Biological: MenABCWY+OMV vaccine
- Naive Group (Experimental): Subjects similar in age to subjects in the MenABCWY+OMV and MenACWY groups, who had not previously received any meningococcal vaccine and who received 2 doses of MenABCWY+OMV vaccine, 1 month apart (Day 1 and Day 31), in the current study.
  Interventions: Biological: MenABCWY+OMV vaccine

INTERVENTIONS:
Biological: MenABCWY+OMV vaccine — Intramuscular injection of a single dose at Day 1 to subjects in the MenABCWY+OMV Group or as a 2 doses at Day 1 and Day 31, one month apart, to subjects in the MenACWY and Naive Groups.

SUMMARY:
The purpose of this study is to evaluate persistence of bactericidal antibodies for N. meningitidis serogroups A, C, W, and Y and serogroup B test strains approximately 4 years after primary vaccination in subjects who previously received a 2-dose series of MenABCWY+Outer membrane Vesicles (OMV) or a single dose of MenACWY, to evaluate immune response against N. meningitidis serogroups A, C, W and Y and serogroup B test strains 30 days after a dose of MenABCWY+OMV in previously vaccinated subjects, and 30 days after a 2-dose series in vaccine-naive subjects of similar age, to evaluate kinetics of immune response at 3, 7, and 30 days after a booster dose of MenABCWY+OMV in previously vaccinated subjects and to explore differences in the kinetics of immune response 3, 7 and 30 days after an accelerated 2 dose series of MenABCWY+OMV separated by 30 days given to vaccine-naive subjects, and to assess immunogenicity of 2 doses of MenABCWY+OMV at Day 61 in vaccine-naive subjects and subjects who previously received one dose of MenACWY

DETAILED DESCRIPTION:
Subjects will be randomised into two different blood draw schedules according to a 1:1 ratio

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who received either 2 doses of MenABCWY+OMV or a single dose of MenACWY followed by a dose of placebo, with the last study vaccine given approximately 48 to 56 months before study V102_02E2 (NCT01367158), who received Tdap only in V102_02E1 (NCT01367158) study and who received no other meningococcal vaccines; Or A proportional number of subjects in each site aged 15 through 23 years on the day of informed consent/assent who did not participate in the V102_02 (NCT01210885) study and have not previously received any meningococcal vaccine.
2. Individuals who / whose parent(s)/legal guardian(s) have voluntarily given written informed consent/assent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Individuals who can comply with study procedures including blood draws and follow-up.
4. Males Or Females of non-childbearing potential Or Females of childbearing potential who are not pregnant or breastfeeding and who are using an effective birth control method which they have used for at least 30 days prior to study entry, and which they intend to use for at least 30 days after the last study vaccination

Exclusion Criteria:

1. History of any meningococcal vaccine administration (study group C) or History of any meningococcal vaccine administration other than vaccination given in the parent V102_02 (NCT01210885) study (study groups A and B).
2. Progressive, unstable or uncontrolled clinical conditions.
3. Hypersensitivity, including allergy, to any component of vac-cines (including diphtheria toxoid (CRM197) and latex) whose use is foreseen in this study.
4. Clinical conditions representing a contraindication to intra-muscular vaccination and blood draws.
5. Abnormal function of the immune system resulting from:

   a.Clinical conditions.
6. Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to enrollment.
7. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
8. Received immunoglobulins or any blood products within 90 days prior to enrollment.
9. Received an investigational or non-registered medicinal product within 30 days prior to enrollment.
10. Received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 14 days from the study vaccines.
11. Study personnel as an immediate family or household member.
12. Who have experienced a moderate or severe acute infection and/or fever (defined as temperature 38°C) within 3 days prior to enrollment.
13. Who have received systemic antibiotic treatment within 3 days prior to enrollment.
14. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.

Ages: 15 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2015-11-14 (Actual); Study Completion 2015-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Santiago, Chile
- GSK Investigational Site, Bogotá, Colombia
- GSK Investigational Site, Panama City, Panama

REFERENCES:
- [Background] Saez-Llorens X, Beltran-Rodriguez J, Novoa Pizarro JM, Mensi I, Keshavan P, Toneatto D. Four-year antibody persistence and response to a booster dose of a pentavalent MenABCWY vaccine administered to healthy adolescents and young adults. Hum Vaccin Immunother. 2018 May 4;14(5):1161-1174. doi: 10.1080/21645515.2018.1457595. Epub 2018 May 9. PMID 29601256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 sites in Panama, 3 sites in Colombia and 1 site in Chile.
Pre-assignment Details: Healthy adolescents and young adults, who received 2 doses of MenABCWY+OMV vaccine or 1 dose of MenACWY in the parent study V102_02 (NCT01210885) and only Tdap vaccination in study V102_02E1 (NCT01367158) were included in the present study along with Naive subjects of similar age.
Period: Overall Study
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Started | 33 | 46 | 50
Completed | 33 | 46 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group | Total
Number analyzed (Participants) | 33 | 46 | 50 | 129
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 18.61 (2.207) | 18.72 (1.87) | 17.96 (2.04) | 18.4 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 25 | 74
  Male | 11 | 19 | 25 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 4 | 3 | 9
  Race: Black or African American | 4 | 2 | 4 | 10
  Race: White | 7 | 6 | 6 | 19
  Race: Other | 20 | 34 | 37 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With hSBA ≥ Lower Limit Quantitation (LLQ) Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: The HT-hSBA assay format was changed in 2015 in response to CBER comments and no new LLQ values were defined as the validation of this format was not relevant. The LLQ cut off values for the old assay format correspond to 8 for serogroups A,C,W and Y and 5 for serogroup B strains and these results are presented in outcome measures 2 and 3 and are considered final in Company's judgement.
Time Frame: At Day 1 (4 years persistence)
Population: Data was not collected for this outcome measure as validation procedure of the hSBA assay was not relevant to the study.
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Percentages of Subjects With hSBA ≥ 8 Against N. Meningitidis Serogroups A, C, W and Y.
Description: Antibody levels against N. meningitidis serogroups A, C, W and Y in subjects who previously received MenABCWY+OMV or MenACWY approximately 4 years earlier, and in Naïve subjects as measured by the percentages of subjects with hSBA ≥ 8.
Time Frame: At Day 1 (4 years persistence)
Population: Analysis was performed on Full Analysis Set immunogenicity persistence population set- all subjects in the enrolled population who provided at least one evaluable serum sample at baseline (visit 1 in this study) and whose assay result was available for at least one strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Percentages of subjects
  Serogroup A | 27 [13.3 to 45.5] | 41 [27.0 to 56.8] | 2 [0.05 to 10.6]
  Serogroup C: number analyzed (Participants) | 32 | 46 | 49
  Serogroup C | 69 [50.0 to 83.9] | 43 [28.9 to 58.9] | 45 [30.7 to 59.8]
  Serogroup W: number analyzed (Participants) | 32 | 46 | 47
  Serogroup W | 75 [56.6 to 88.5] | 78 [63.6 to 89.1] | 53 [38.1 to 67.9]
  Serogroup Y: number analyzed (Participants) | 32 | 44 | 47
  Serogroup Y | 38 [21.1 to 56.3] | 59 [43.2 to 73.7] | 19 [9.1 to 33.3]

3. Primary Outcome: Percentages of Subjects With hSBA ≥ 5 Against N. Meningitidis Serogroup B Test Strains.
Description: Antibody levels against N. meningitidis serogroup B test strains in subjects who previously received MenABCWY+OMV or MenACWY approximately 4 years earlier, and in Naïve subjects as measured by the percentages of Subjects with hSBA ≥ 5. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Day 1 (4 years persistence)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Percentages of subjects
  Serogroup B, M14459 | 18 [7.0 to 35.5] | 4 [0.5 to 14.8] | 8 [2.2 to 19.2]
  Serogroup B, M01-0240364: number analyzed (Participants) | 31 | 44 | 50
  Serogroup B, M01-0240364 | 13 [3.6 to 29.8] | 5 [0.6 to 15.5] | 4 [0.49 to 13.7]
  Serogroup B, NZ98/254 | 15 [5.1 to 31.9] | 2 [0.06 to 11.5] | 6 [1.3 to 16.5]
  Serogroup B, M10713 | 48 [30.8 to 66.5] | 33 [19.5 to 48.0] | 38 [24.7 to 52.8]
  Serogroup B, H44/76 | 27 [13.3 to 45.5] | 4 [0.5 to 14.8] | 10 [3.3 to 21.8]
  Serogroup B, 5/99 | 70 [51.3 to 84.4] | 17 [7.8 to 31.4] | 16 [7.2 to 29.1]

4. Primary Outcome: Geometric Mean hSBA Titers (GMTs) Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMTs against N. meningitidis serogroups A, C, W and Y and serogroup B test strains in subjects who previously received MenABCWY+OMV or MenACWY approximately 4 years earlier, and in Naïve subjects. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Titers
  Serogroup B, M14459 | 2.04 [1.46 to 2.83] | 1.37 [1.12 to 1.69] | 1.48 [1.18 to 1.85]
  Serogroup B, M01-0240364: number analyzed (Participants) | 31 | 44 | 50
  Serogroup B, M01-0240364 | 2.26 [1.26 to 4.08] | 1.14 [0.97 to 1.35] | 1.23 [1.02 to 1.47]
  Serogroup B, NZ98/254 | 1.81 [1.30 to 2.51] | 1.35 [1.15 to 1.59] | 1.45 [1.18 to 1.77]
  Serogroup B, M10713 | 3.66 [2.38 to 5.62] | 2.56 [1.74 to 3.75] | 3.10 [2.16 to 4.45]
  Serogroup B, H44/76 | 2.33 [1.57 to 3.45] | 1.21 [1.03 to 1.42] | 1.44 [1.14 to 1.80]
  Serogroup B, 5/99 | 13 [7.29 to 22] | 1.78 [1.36 to 2.34] | 1.90 [1.42 to 2.53]
  Serogroup A | 4.06 [2.22 to 7.44] | 6.64 [3.56 to 12] | 1.20 [1.05 to 1.37]
  Serogroup C: number analyzed (Participants) | 32 | 46 | 49
  Serogroup C | 17 [7.80 to 37] | 6.62 [4.10 to 11] | 5.11 [3.49 to 7.48]
  Serogroup W: number analyzed (Participants) | 32 | 46 | 47
  Serogroup W | 28 [15 to 53] | 25 [15 to 40] | 8.37 [4.78 to 15]
  Serogroup Y: number analyzed (Participants) | 32 | 44 | 47
  Serogroup Y | 6.17 [3.00 to 13] | 12 [6.29 to 22] | 2.00 [1.40 to 2.85]
Statistical Analysis 1: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M14459; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.48, 95% CI 2-sided [1.03 to 2.12]
Statistical Analysis 2: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M14459; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.93, 95% CI 2-sided [0.67 to 1.28]
Statistical Analysis 3: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M14459; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.38, 95% CI 2-sided [0.97 to 1.96]
Statistical Analysis 4: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M01-0240364; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.98, 95% CI 2-sided [1.27 to 3.09]
Statistical Analysis 5: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M01-0240364; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.93, 95% CI 2-sided [0.63 to 1.37]
Statistical Analysis 6: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M01-0240364; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.84, 95% CI 2-sided [1.20 to 2.84]
Statistical Analysis 7: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, NZ98/254; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.34, 95% CI 2-sided [0.96 to 1.85]
Statistical Analysis 8: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, NZ98/254; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.94, 95% CI 2-sided [0.70 to 1.25]
Statistical Analysis 9: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, NZ98/254; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.25, 95% CI 2-sided [0.91 to 1.72]
Statistical Analysis 10: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M10713; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.43, 95% CI 2-sided [0.81 to 2.53]
Statistical Analysis 11: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M10713; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.82, 95% CI 2-sided [0.49 to 1.37]
Statistical Analysis 12: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M10713; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.18, 95% CI 2-sided [0.67 to 2.06]
Statistical Analysis 13: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, H44/76; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.92, 95% CI 2-sided [1.33 to 2.78]
Statistical Analysis 14: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, H44/76; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.84, 95% CI 2-sided [0.61 to 1.17]
Statistical Analysis 15: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, H44/76; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.62, 95% CI 2-sided [1.13 to 2.32]
Statistical Analysis 16: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, 5/99; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 7.15, 95% CI 2-sided [4.25 to 12]
Statistical Analysis 17: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, 5/99; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.94, 95% CI 2-sided [0.59 to 1.50]
Statistical Analysis 18: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, 5/99; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 6.73, 95% CI 2-sided [4.03 to 11]
Statistical Analysis 19: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup A; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.61, 95% CI 2-sided [0.30 to 1.23]
Statistical Analysis 20: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup A; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 5.53, 95% CI 2-sided [2.96 to 10]
Statistical Analysis 21: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup A; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 3.38, 95% CI 2-sided [1.70 to 6.73]
Statistical Analysis 22: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup C; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 2.58, 95% CI 2-sided [1.20 to 5.54]
Statistical Analysis 23: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup C; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.30, 95% CI 2-sided [0.66 to 2.56]
Statistical Analysis 24: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup C; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 3.34, 95% CI 2-sided [1.57 to 7.11]
Statistical Analysis 25: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup W; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.14, 95% CI 2-sided [0.51 to 2.59]
Statistical Analysis 26: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup W; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 2.93, 95% CI 2-sided [1.40 to 6.12]
Statistical Analysis 27: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup W; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 3.35, 95% CI 2-sided [1.49 to 7.57]
Statistical Analysis 28: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup Y; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.52, 95% CI 2-sided [0.23 to 1.18]
Statistical Analysis 29: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup Y; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 5.94, 95% CI 2-sided [2.84 to 12]
Statistical Analysis 30: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup Y; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 3.09, 95% CI 2-sided [1.38 to 6.92]

5. Primary Outcome: Percentages of Subjects With hSBA ≥ LLQ Against N. Meningitidis Serogroups A, C, W and Y and B Test Strains.
Description: The HT-hSBA assay format was changed in 2015 in response to CBER comments and no new LLQ values were defined as the validation of this format was not relevant. The LLQ cut off values for the old assay format correspond to 8 for serogroups A,C,W and Y and 5 for serogroup B strains and these results are presented in outcome measures 6 and 7 and are considered final in Company's judgement.
Time Frame: At Day 31
Population: Data was not collected for this outcome measure as validation procedure of the hSBA assay was not relevant to the study.
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Percentages of Subjects With hSBA ≥ 8 Against N. Meningitidis Serogroups A, C, W and Y.
Description: Immune response against N. meningitidis serogroups A, C, W and Y 30 days after a single dose of MenABCWY+OMV in subjects who previously vaccinated subjects, and in Naïve subjects of similar age, as measured by the percentages of subjects with hSBA ≥ 8.
Time Frame: At Day 31
Population: Analysis was performed on Full Analysis Set immunogenicity persistence population set Day 31- all subjects in the enrolled population who received a study vaccination, provided at least one evaluable serum sample at 1 month post vaccination and whose assay result was available for at least one strain.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Percentage of Subjects
  Serogroup A | 100 [89.4 to 100.0] | 100 [92.3 to 100.0] | 76 [61.8 to 86.9]
  Serogroup C: number analyzed (Participants) | 30 | 38 | 48
  Serogroup C | 100 [88.4 to 100.0] | 100 [90.7 to 100.0] | 94 [82.8 to 98.7]
  Serogroup W: number analyzed (Participants) | 28 | 38 | 46
  Serogroup W | 100 [87.7 to 100.0] | 100 [90.7 to 100.0] | 96 [85.2 to 99.5]
  Serogroup Y: number analyzed (Participants) | 23 | 23 | 46
  Serogroup Y | 100 [85.2 to 100.0] | 100 [85.2 to 100.0] | 85 [71.1 to 93.7]

7. Primary Outcome: Percentages of Subjects With hSBA ≥ 5 Against N. Meningitidis Serogroup B Test Strains.
Description: Immune response against N. meningitidis serogroup B test strains 30 days after a single dose of MenABCWY+OMV in previously vaccinated subjects, and in Naïve subjects of similar age, as measured by the percentages of Subjects with hSBA ≥ 5. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Day 31
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Percentages of Subjects
  Serogroup B, M14459: number analyzed (Participants) | 33 | 45 | 50
  Serogroup B, M14459 | 85 [68.1 to 94.9] | 31 [18.2 to 46.6] | 40 [26.4 to 54.8]
  Serogroup B, M01-0240364: number analyzed (Participants) | 30 | 44 | 45
  Serogroup B, M01-0240364 | 97 [82.8 to 99.92] | 25 [13.2 to 40.3] | 29 [16.4 to 44.3]
  Serogroup B, NZ98/254 | 82 [64.5 to 93.0] | 37 [23.2 to 52.5] | 52 [37.4 to 66.3]
  Serogroup B, M10713 | 85 [68.1 to 94.9] | 52 [36.9 to 67.1] | 58 [43.2 to 71.8]
  Serogroup B, H44/76 | 97 [84.2 to 99.92] | 52 [36.9 to 67.1] | 60 [45.2 to 73.6]
  Serogroup B, 5/99 | 100 [89.4 to 100.0] | 78 [63.6 to 89.1] | 82 [68.6 to 91.4]

8. Primary Outcome: Geometric Mean hSBA Titers (GMTs) Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMTs against N. meningitidis serogroups A, C, W and Y and serogroup B test strains 30 days after a single dose of MenABCWY+OMV in previously vaccinated subjects, and in Naïve subjects of similar age. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Day 31
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Titers
  Serogroup B, M14459: number analyzed (Participants) | 33 | 45 | 50
  Serogroup B, M14459 | 24 [14 to 42] | 2.83 [1.88 to 4.24] | 4.02 [2.67 to 6.06]
  Serogroup B, M01-0240364: number analyzed (Participants) | 30 | 44 | 45
  Serogroup B, M01-0240364 | 601 [339 to 1064] | 3.05 [1.77 to 5.26] | 3.11 [1.76 to 5.51]
  Serogroup B, NZ98/254 | 13 [8.50 to 18] | 3.57 [2.37 to 5.38] | 5.75 [3.95 to 8.37]
  Serogroup B, M10713 | 20 [13 to 31] | 5.51 [3.45 to 8.79] | 7.70 [5.04 to 12]
  Serogroup B, H44/76 | 98 [57 to 170] | 5.78 [3.59 to 9.31] | 7.27 [4.53 to 12]
  Serogroup B, 5/99 | 1426 [940 to 2164] | 19 [11 to 34] | 25 [15 to 42]
  Serogroup A | 396 [288 to 545] | 149 [106 to 210] | 22 [14 to 35]
  Serogroup C: number analyzed (Participants) | 30 | 38 | 48
  Serogroup C | 1676 [1164 to 2414] | 1199 [849 to 1692] | 58 [35 to 96]
  Serogroup W: number analyzed (Participants) | 28 | 38 | 46
  Serogroup W | 1823 [1163 to 2856] | 2259 [1678 to 3041] | 117 [83 to 166]
  Serogroup Y: number analyzed (Participants) | 23 | 23 | 46
  Serogroup Y | 779 [430 to 1413] | 1692 [1206 to 2373] | 85 [45 to 163]
Statistical Analysis 1: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M14459; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 8.50, 95% CI 2-sided [4.41 to 16]
Statistical Analysis 2: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M14459; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.70, 95% CI 2-sided [0.39 to 1.27]
Statistical Analysis 3: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M14459; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 5.97, 95% CI 2-sided [3.14 to 11]
Statistical Analysis 4: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M01-0240364; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 197, 95% CI 2-sided [86 to 452]
Statistical Analysis 5: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M01-0240364; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.98, 95% CI 2-sided [0.47 to 2.07]
Statistical Analysis 6: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M01-0240364; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 193, 95% CI 2-sided [84 to 442]
Statistical Analysis 7: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, NZ98/254; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 3.51, 95% CI 2-sided [1.96 to 6.27]
Statistical Analysis 8: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, NZ98/254; Test type: Other; Mixed Models Analysis; Geometric mean ratio = 0.62, 95% CI 2-sided [0.37 to 1.0]
Statistical Analysis 9: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, NZ98/254; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 2.17, 95% CI 2-sided [1.23 to 3.85]
Statistical Analysis 10: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M10713; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 3.57, 95% CI 2-sided [1.84 to 6.92]
Statistical Analysis 11: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M10713; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.72, 95% CI 2-sided [0.40 to 1.29]
Statistical Analysis 12: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, M10713; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 2.55, 95% CI 2-sided [1.33 to 4.89]
Statistical Analysis 13: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, H44/76; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 17, 95% CI 2-sided [8.18 to 35]
Statistical Analysis 14: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, H44/76; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.80, 95% CI 2-sided [0.41 to 1.53]
Statistical Analysis 15: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, H44/76; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 13, 95% CI 2-sided [6.59 to 28]
Statistical Analysis 16: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, 5/99; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 74, 95% CI 2-sided [34 to 160]
Statistical Analysis 17: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, 5/99; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.77, 95% CI 2-sided [0.38 to 1.53]
Statistical Analysis 18: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B, 5/99; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 57, 95% CI 2-sided [27 to 121]
Statistical Analysis 19: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup A; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 2.66, 95% CI 2-sided [1.46 to 4.83]
Statistical Analysis 20: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup A; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 6.76, 95% CI 2-sided [3.96 to 12]
Statistical Analysis 21: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup A; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 18, 95% CI 2-sided [10 to 32]
Statistical Analysis 22: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup C; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 1.40, 95% CI 2-sided [0.72 to 2.71]
Statistical Analysis 23: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup C; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 21, 95% CI 2-sided [12 to 37]
Statistical Analysis 24: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup C; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 29, 95% CI 2-sided [15 to 55]
Statistical Analysis 25: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup W; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.81, 95% CI 2-sided [0.47 to 1.38]
Statistical Analysis 26: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup W; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 19, 95% CI 2-sided [12 to 31]
Statistical Analysis 27: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup W; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 16, 95% CI 2-sided [9.27 to 26]
Statistical Analysis 28: Comparison: MenABCWY+OMV Group vs MenACWY Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup Y; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.46, 95% CI 2-sided [0.17 to 1.28]
Statistical Analysis 29: Comparison: MenACWY Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup Y; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 20, 95% CI 2-sided [8.20 to 48]
Statistical Analysis 30: Comparison: MenABCWY+OMV Group vs Naive Group; Between-group Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup Y; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 9.13, 95% CI 2-sided [3.78 to 22]

9. Primary Outcome: Geometric Mean hSBA Ratio (GMRs) Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMRs as measure of the immune response against N. meningitidis serogroups A, C, W and Y and serogroup B test strains in previously vaccinated subjects, and in Naïve subjects of similar age. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: Day 31 versus Day 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Ratios
  Serogroup B, M14459: number analyzed (Participants) | 33 | 45 | 50
  Serogroup B, M14459 | 12 [6.88 to 20] | 2.11 [1.45 to 3.07] | 2.72 [1.91 to 3.87]
  Serogroup B, M01-0240364: number analyzed (Participants) | 28 | 42 | 45
  Serogroup B, M01-0240364 | 229 [108 to 485] | 2.80 [1.59 to 4.96] | 2.48 [1.51 to 4.07]
  Serogroup B, NZ98/254 | 6.92 [4.61 to 10] | 2.64 [1.73 to 4.02] | 3.98 [2.73 to 5.79]
  Serogroup B, M10713 | 5.38 [3.54 to 8.17] | 2.15 [1.46 to 3.17] | 2.48 [1.78 to 3.45]
  Serogroup B, H44/76 | 42 [25 to 72] | 4.78 [2.90 to 7.89] | 5.06 [3.21 to 7.97]
  Serogroup B, 5/99 | 112 [68 to 185] | 11 [6.09 to 19] | 13 [8.14 to 22]
  Serogroup A | 98 [54 to 177] | 22 [13 to 38] | 18 [12 to 29]
  Serogroup C: number analyzed (Participants) | 30 | 38 | 48
  Serogroup C | 105 [49 to 222] | 238 [145 to 392] | 12 [6.88 to 19]
  Serogroup W: number analyzed (Participants) | 28 | 38 | 44
  Serogroup W | 67 [34 to 132] | 112 [65 to 191] | 16 [8.35 to 30]
  Serogroup Y: number analyzed (Participants) | 22 | 22 | 23
  Serogroup Y | 162 [70 to 375] | 216 [80 to 580] | 46 [23 to 92]

10. Secondary Outcome: Percentages of Subjects With hSBA ≥ LLQ Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: The HT-hSBA assay format was changed in 2015 in response to CBER comments and no new LLQ values were defined as the validation of this format was not relevant. The LLQ cut off values for the old assay format correspond to 8 for serogroups A,C,W and Y and 5 for serogroup B strains and these results are presented in outcome measures 12 and 13 and are considered final in Company's judgement.
Time Frame: At Days 1, 4, 8 and 31
Population: Data was not collected for this outcome measure as validation procedure of the hSBA assay was not relevant to the study.
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Percentages of Subjects With hSBA ≥ LLQ Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: as for outcome 10
Time Frame: At Days 1, 31, 34, 38 and 61
Population: Data was not collected for this outcome measure as validation procedure of the hSBA assay was not relevant to the study.
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Percentages of Subjects With hSBA ≥ 8 Against N. Meningitidis Serogroups A, C, W and Y.
Description: Kinetics of immune response following 1 dose of MenABCWY+OMV in subjects who previously received 2 doses of MenABCWY+OMV or 1 dose of MenACWY, at Days 1, 4, 8, 31, 34, 38 and 61, as measured by the percentages of subjects with hSBA ≥ 8.
Time Frame: At Days 1, 4, 8, 31, 34, 38 and 61
Population: Analysis was performed on Full Analysis Set immunogenicity kinetics population set- all subjects in the enrolled population who received a study vaccination, provided at least one evaluable serum sample post vaccination and whose assay result was available for at least one strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenABCWY+OMV Group (A): Subjects who received 2 doses of MenABCWY+OMV vaccine in the parent study V102_02 (NCT01210885) and received no subsequent meningococcal vaccines, received a booster dose of MenABCWY+OMV vaccine in the current study at Day 1. Blood samples will be collected from subjects at Day 1 (before vaccination), Day 4, Day 8 and Day 31.
- MenACWY Group (B1): Subjects who received MenACWY vaccine in the parent study V102_02 (NCT01210885) and received no subsequent meningococcal vaccines, received 2 doses of MenABCWY+OMV vaccine, one month apart, in the current study. Blood samples will be collected from subjects at Day 1 (before vaccination), Day 4, Day 31 (before vaccination) and Day 61.
- MenACWY Group (B2): Subjects who received MenACWY vaccine in the parent study V102_02 (NCT01210885) and received no subsequent meningococcal vaccines, received 2 doses of MenABCWY+OMV vaccine, one month apart, in the current study. Blood samples will be collected from subjects at Day 1 (before vaccination), Day 8, Day 31 (before vaccination) and Day 61.
- Naive Group (C1): Subjects similar in age to subjects in the MenABCWY+OMV and MenACWY groups, who had not previously received any meningococcal vaccine and who received 2 doses of MenABCWY+OMV vaccine, 1 month apart (Day 1 and Day 31), in the current study. Blood samples will be collected from subjects at Day 1 (before vaccination), Day 31 (before vaccination), Day 34 and Day 61.
- Naive Group (C2): Subjects similar in age to subjects in the MenABCWY+OMV and MenACWY groups, who had not previously received any meningococcal vaccine and who received 2 doses of MenABCWY+OMV vaccine, 1 month apart (Day 1 and Day 31), in the current study. Blood samples will be collected from subjects at Day 1 (before vaccination), Day 31 (before vaccination), Day 38 and Day 61.
Arm/Group | MenABCWY+OMV Group (A) | MenACWY Group (B1) | MenACWY Group (B2) | Naive Group (C1) | Naive Group (C2)
Number analyzed (Participants) | 33 | 23 | 23 | 26 | 24
Percentages of subjects
  Serogroup A; Day 1 | 27 [13.3 to 45.5] | 52 [30.6 to 73.2] | 30 [13.2 to 52.9] | 0 [0.0 to 13.2] | 4 [0.11 to 21.1]
  Serogroup A; Day 4: number analyzed (Participants) | 33 | 23 | 0 | 0 | 0
  Serogroup A; Day 4 | 24 [11.1 to 42.3] | 52 [30.6 to 73.2] |  |  |
  Serogroup A; Day 8: number analyzed (Participants) | 33 | 0 | 22 | 0 | 0
  Serogroup A; Day 8 | 100 [89.4 to 100.0] |  | 82 [59.7 to 94.8] |  |
  Serogroup A; Day 31 | 100 [89.4 to 100.0] | 100 [85.2 to 100.0] | 100 [85.2 to 100.0] | 73 [52.2 to 88.4] | 79 [57.8 to 92.9]
  Serogroup A; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 26 | 0
  Serogroup A; Day 34 |  |  |  | 77 [56.4 to 91.0] |
  Serogroup A; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24
  Serogroup A; Day 38 |  |  |  |  | 96 [78.9 to 99.89]
  Serogroup A; Day 61: number analyzed (Participants) | 0 | 23 | 23 | 23 | 24
  Serogroup A; Day 61 |  | 100 [85.2 to 100.0] | 100 [85.2 to 100.0] | 100 [85.2 to 100.0] | 88 [67.6 to 97.3]
  Serogroup C; Day 1: number analyzed (Participants) | 32 | 23 | 23 | 25 | 24
  Serogroup C; Day 1 | 69 [50.0 to 83.9] | 61 [38.5 to 80.3] | 26 [10.2 to 48.4] | 40 [21.1 to 61.3] | 50 [29.1 to 70.9]
  Serogroup C; Day 4: number analyzed (Participants) | 30 | 22 | 0 | 0 | 0
  Serogroup C; Day 4 | 73 [54.1 to 87.7] | 64 [40.7 to 82.8] |  |  |
  Serogroup C; Day 8: number analyzed (Participants) | 29 | 0 | 19 | 0 | 0
  Serogroup C; Day 8 | 100 [88.1 to 100.0] |  | 100 [82.4 to 100.0] |  |
  Serogroup C; Day 31: number analyzed (Participants) | 30 | 17 | 21 | 25 | 23
  Serogroup C; Day 31 | 100 [88.4 to 100.0] | 100 [80.5 to 100.0] | 100 [83.9 to 100.0] | 100 [86.3 to 100.0] | 87 [66.4 to 97.2]
  Serogroup C; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 20 | 0
  Serogroup C; Day 34 |  |  |  | 100 [83.2 to 100.0] |
  Serogroup C; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 22
  Serogroup C; Day 38 |  |  |  |  | 100 [84.6 to 100.0]
  Serogroup C; Day 61: number analyzed (Participants) | 0 | 15 | 19 | 24 | 23
  Serogroup C; Day 61 |  | 100 [78.2 to 100.0] | 100 [82.4 to 100.0] | 100 [85.8 to 100.0] | 100 [85.2 to 100.0]
  Serogroup W; Day 1: number analyzed (Participants) | 32 | 23 | 23 | 25 | 22
  Serogroup W; Day 1 | 75 [56.6 to 88.5] | 70 [47.1 to 86.8] | 87 [66.4 to 97.2] | 44 [24.4 to 65.1] | 64 [40.7 to 82.8]
  Serogroup W; Day 4: number analyzed (Participants) | 25 | 22 | 0 | 0 | 0
  Serogroup W; Day 4 | 76 [54.9 to 90.6] | 73 [49.8 to 89.3] |  |  |
  Serogroup W; Day 8: number analyzed (Participants) | 25 | 0 | 16 | 0 | 0
  Serogroup W; Day 8 | 100 [86.3 to 100.0] |  | 100 [79.4 to 100.0] |  |
  Serogroup W; Day 31: number analyzed (Participants) | 28 | 17 | 21 | 22 | 24
  Serogroup W; Day 31 | 100 [87.7 to 100.0] | 100 [80.5 to 100.0] | 100 [83.9 to 100.0] | 100 [84.6 to 100.0] | 92 [73.0 to 99.0]
  Serogroup W; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 19 | 0
  Serogroup W; Day 34 |  |  |  | 100 [82.4 to 100.0] |
  Serogroup W; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 20
  Serogroup W; Day 38 |  |  |  |  | 100 [83.2 to 100.0]
  Serogroup W; Day 61: number analyzed (Participants) | 0 | 15 | 17 | 20 | 21
  Serogroup W; Day 61 |  | 100 [78.2 to 100.0] | 100 [80.5 to 100.0] | 100 [83.2 to 100.0] | 100 [83.9 to 100.0]
  Serogroup Y; Day 1: number analyzed (Participants) | 32 | 22 | 22 | 23 | 24
  Serogroup Y; Day 1 | 38 [21.1 to 56.3] | 64 [40.7 to 82.8] | 55 [32.2 to 75.6] | 17 [5.0 to 38.8] | 21 [7.1 to 42.2]
  Serogroup Y; Day 4: number analyzed (Participants) | 31 | 22 | 0 | 0 | 0
  Serogroup Y; Day 4 | 42 [24.5 to 60.9] | 50 [28.2 to 71.8] |  |  |
  Serogroup Y; Day 8: number analyzed (Participants) | 23 | 0 | 13 | 0 | 0
  Serogroup Y; Day 8 | 100 [85.2 to 100.0] |  | 100 [75.3 to 100.0] |  |
  Serogroup Y; Day 31: number analyzed (Participants) | 23 | 12 | 11 | 23 | 23
  Serogroup Y; Day 31 | 100 [85.2 to 100.0] | 100 [73.5 to 100.0] | 100 [71.5 to 100.0] | 91 [72.0 to 98.9] | 78 [56.3 to 92.5]
  Serogroup Y; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 23 | 0
  Serogroup Y; Day 34 |  |  |  | 96 [78.1 to 99.89] |
  Serogroup Y; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 20
  Serogroup Y; Day 38 |  |  |  |  | 100 [83.2 to 100.0]
  Serogroup Y; Day 61: number analyzed (Participants) | 0 | 12 | 15 | 23 | 20
  Serogroup Y; Day 61 |  | 100 [73.5 to 100.0] | 100 [78.2 to 100.0] | 100 [85.2 to 100.0] | 95 [75.1 to 99.87]

13. Secondary Outcome: Percentages of Subjects With hSBA ≥ 5 Against N. Meningitidis Serogroup B Test Strains.
Description: Kinetics of immune response against N. meningitidis serogroup B test strains in previously vaccinated subjects, at Days 1, 4, 8, 31, 34, 38 and 61, as measured by the percentages of Subjects with hSBA ≥ 5. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Days 1, 4, 8, 31, 34, 38 and 61
Population: Kinetics of immune response against N. meningitidis serogroup B test strains in previously vaccinated subjects, at Day 1, 4, 8, 31, as measured by the percentages of Subjects with hSBA ≥ 5. The data were reported based on the FAS immunogenicity kinetics population set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY+OMV Group (A) | MenACWY Group (B1) | MenACWY Group (B2) | Naive Group (C1) | Naive Group (C2)
Number analyzed (Participants) | 33 | 23 | 23 | 26 | 24
Percentages of subjects
  Serogroup B, M14459; Day 1 | 18 [7.0 to 35.5] | 9 [1.1 to 28.0] | 0 [0.0 to 14.8] | 8 [0.9 to 25.1] | 8 [1.0 to 27.0]
  Serogroup B, M14459; Day 4: number analyzed (Participants) | 33 | 23 | 0 | 0 | 0
  Serogroup B, M14459; Day 4 | 21 [9.0 to 38.9] | 4 [0.11 to 21.9] |  |  |
  Serogroup B, M14459; Day 8: number analyzed (Participants) | 33 | 0 | 22 | 0 | 0
  Serogroup B, M14459; Day 8 | 79 [61.1 to 91.0] |  | 14 [2.9 to 34.9] |  |
  Serogroup B, M14459; Day 31: number analyzed (Participants) | 33 | 23 | 22 | 26 | 24
  Serogroup B, M14459; Day 31 | 85 [68.1 to 94.9] | 35 [16.4 to 57.3] | 27 [10.7 to 50.2] | 46 [26.6 to 66.6] | 33 [15.6 to 55.3]
  Serogroup B, M14459; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 26 | 0
  Serogroup B, M14459; Day 34 |  |  |  | 42 [23.4 to 63.1] |
  Serogroup B, M14459; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24
  Serogroup B, M14459; Day 38 |  |  |  |  | 71 [48.9 to 87.4]
  Serogroup B, M14459; Day 61: number analyzed (Participants) | 0 | 23 | 23 | 25 | 24
  Serogroup B, M14459; Day 61 |  | 43 [23.2 to 65.5] | 48 [26.8 to 69.4] | 80 [59.3 to 93.2] | 54 [32.8 to 74.4]
  Serogroup B, M01-0240364; Day 1: number analyzed (Participants) | 31 | 22 | 22 | 26 | 24
  Serogroup B, M01-0240364; Day 1 | 13 [3.6 to 29.8] | 9 [1.1 to 29.2] | 0 [0.0 to 15.4] | 4 [0.10 to 19.6] | 4 [0.11 to 21.1]
  Serogroup B, M01-0240364; Day 4: number analyzed (Participants) | 30 | 23 | 0 | 0 | 0
  Serogroup B, M01-0240364; Day 4 | 17 [5.6 to 34.7] | 4 [0.11 to 21.9] |  |  |
  Serogroup B, M01-0240364; Day 8: number analyzed (Participants) | 29 | 0 | 21 | 0 | 0
  Serogroup B, M01-0240364; Day 8 | 93 [77.2 to 99.2] |  | 10 [1.2 to 30.4] |  |
  Serogroup B, M01-0240364; Day 31: number analyzed (Participants) | 30 | 21 | 23 | 24 | 21
  Serogroup B, M01-0240364; Day 31 | 97 [82.8 to 99.92] | 29 [11.3 to 52.2] | 22 [7.5 to 43.7] | 33 [15.6 to 55.3] | 24 [8.2 to 47.2]
  Serogroup B, M01-0240364; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 25 | 0
  Serogroup B, M01-0240364; Day 34 |  |  |  | 40 [21.1 to 61.3] |
  Serogroup B, M01-0240364; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 22
  Serogroup B, M01-0240364; Day 38 |  |  |  |  | 82 [59.7 to 94.8]
  Serogroup B, M01-0240364; Day 61: number analyzed (Participants) | 0 | 23 | 23 | 23 | 24
  Serogroup B, M01-0240364; Day 61 |  | 65 [42.7 to 83.6] | 65 [42.7 to 83.6] | 70 [47.1 to 86.8] | 71 [48.9 to 87.4]
  Serogroup B, NZ98/254; Day 1 | 15 [5.1 to 31.9] | 4 [0.11 to 21.9] | 0 [0.0 to 14.8] | 8 [0.9 to 25.1] | 4 [0.11 to 21.1]
  Serogroup B, NZ98/254; Day 4: number analyzed (Participants) | 33 | 23 | 0 | 0 | 0
  Serogroup B, NZ98/254; Day 4 | 12 [3.4 to 28.2] | 13 [2.8 to 33.6] |  |  |
  Serogroup B, NZ98/254; Day 8: number analyzed (Participants) | 33 | 0 | 22 | 0 | 0
  Serogroup B, NZ98/254; Day 8 | 67 [48.2 to 82.0] |  | 9 [1.1 to 29.2] |  |
  Serogroup B, NZ98/254; Day 31 | 82 [64.5 to 93.0] | 48 [26.8 to 69.4] | 26 [10.2 to 48.4] | 58 [36.9 to 76.6] | 46 [25.6 to 67.2]
  Serogroup B, NZ98/254; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 26 | 0
  Serogroup B, NZ98/254; Day 34 |  |  |  | 50 [29.9 to 70.1] |
  Serogroup B, NZ98/254; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24
  Serogroup B, NZ98/254; Day 38 |  |  |  |  | 75 [53.3 to 90.2]
  Serogroup B, NZ98/254; Day 61: number analyzed (Participants) | 0 | 23 | 23 | 25 | 24
  Serogroup B, NZ98/254; Day 61 |  | 52 [30.6 to 73.2] | 39 [19.7 to 61.5] | 72 [50.6 to 87.9] | 50 [29.1 to 70.9]
  Serogroup B, M10713; Day 1 | 48 [30.8 to 66.5] | 48 [26.8 to 69.4] | 17 [5.0 to 38.8] | 38 [20.2 to 59.4] | 38 [18.8 to 59.4]
  Serogroup B, M10713; Day 4: number analyzed (Participants) | 32 | 23 | 0 | 0 | 0
  Serogroup B, M10713; Day 4 | 56 [37.7 to 73.6] | 39 [19.7 to 61.5] |  |  |
  Serogroup B, M10713; Day 8: number analyzed (Participants) | 33 | 0 | 22 | 0 | 0
  Serogroup B, M10713; Day 8 | 79 [61.1 to 91.0] |  | 32 [13.9 to 54.9] |  |
  Serogroup B, M10713; Day 31 | 85 [68.1 to 94.9] | 70 [47.1 to 86.8] | 35 [16.4 to 57.3] | 62 [40.6 to 79.8] | 54 [32.8 to 74.4]
  Serogroup B, M10713; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 23 | 0
  Serogroup B, M10713; Day 34 |  |  |  | 57 [34.5 to 76.8] |
  Serogroup B, M10713; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24
  Serogroup B, M10713; Day 38 |  |  |  |  | 67 [44.7 to 84.4]
  Serogroup B, M10713; Day 61: number analyzed (Participants) | 0 | 23 | 23 | 25 | 24
  Serogroup B, M10713; Day 61 |  | 65 [42.7 to 83.6] | 43 [23.2 to 65.5] | 68 [46.5 to 85.1] | 63 [40.6 to 81.2]
  Serogroup B, H44/76; Day 1 | 27 [13.3 to 45.5] | 9 [1.1 to 28.0] | 0 [0.0 to 14.8] | 12 [2.4 to 30.2] | 8 [1.0 to 27.0]
  Serogroup B, H44/76; Day 4: number analyzed (Participants) | 33 | 23 | 0 | 0 | 0
  Serogroup B, H44/76; Day 4 | 21 [9.0 to 38.9] | 4 [0.11 to 21.9] |  |  |
  Serogroup B, H44/76; Day 8: number analyzed (Participants) | 33 | 0 | 22 | 0 | 0
  Serogroup B, H44/76; Day 8 | 94 [79.8 to 99.3] |  | 14 [2.9 to 34.9] |  |
  Serogroup B, H44/76; Day 31 | 97 [84.2 to 99.92] | 52 [30.6 to 73.2] | 52 [30.6 to 73.2] | 73 [52.2 to 88.4] | 46 [25.6 to 67.2]
  Serogroup B, H44/76; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 26 | 0
  Serogroup B, H44/76; Day 34 |  |  |  | 69 [48.2 to 85.7] |
  Serogroup B, H44/76; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24
  Serogroup B, H44/76; Day 38 |  |  |  |  | 96 [78.9 to 99.89]
  Serogroup B, H44/76; Day 61: number analyzed (Participants) | 0 | 23 | 23 | 25 | 24
  Serogroup B, H44/76; Day 61 |  | 78 [56.3 to 92.5] | 91 [72.0 to 98.9] | 96 [79.6 to 99.90] | 79 [57.8 to 92.9]
  Serogroup B, 5/99; Day 1 | 70 [51.3 to 84.4] | 22 [7.5 to 43.7] | 13 [2.8 to 33.6] | 19 [6.6 to 39.4] | 13 [2.7 to 32.4]
  Serogroup B, 5/99; Day 4: number analyzed (Participants) | 33 | 23 | 0 | 0 | 0
  Serogroup B, 5/99; Day 4 | 79 [61.1 to 91.0] | 9 [1.1 to 28.0] |  |  |
  Serogroup B, 5/99; Day 8: number analyzed (Participants) | 33 | 0 | 22 | 0 | 0
  Serogroup B, 5/99; Day 8 | 100 [89.4 to 100.0] |  | 9 [1.1 to 29.2] |  |
  Serogroup B, 5/99; Day 31 | 100 [89.4 to 100.0] | 78 [56.3 to 92.5] | 78 [56.3 to 92.5] | 85 [65.1 to 95.6] | 79 [57.8 to 92.9]
  Serogroup B, 5/99; Day 34: number analyzed (Participants) | 0 | 0 | 0 | 26 | 0
  Serogroup B, 5/99; Day 34 |  |  |  | 85 [65.1 to 95.6] |
  Serogroup B, 5/99; Day 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24
  Serogroup B, 5/99; Day 38 |  |  |  |  | 100 [85.8 to 100.0]
  Serogroup B, 5/99; Day 61: number analyzed (Participants) | 0 | 23 | 23 | 25 | 24
  Serogroup B, 5/99; Day 61 |  | 100 [85.2 to 100.0] | 100 [85.2 to 100.0] | 100 [86.3 to 100.0] | 100 [85.8 to 100.0]

14. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMTs at Day 1, 4, 8, 31 as measure of the kinetics of the immune response following a dose of MenABCWY+OMV, in subjects who previously received 2 doses of MenABCWY+OMV or 1 dose of MenACWY. This outcome measure reports data only for the MenABCWY+OMV and MenACWY Groups as per protocol. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Days 1, 4, 8 and 31.
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY+OMV Group | MenACWY Group
Number analyzed (Participants) | 33 | 46
Titers
  Serogroup B, M14459; Day 1 | 2.04 [1.46 to 2.83] | 1.37 [1.12 to 1.69]
  Serogroup B, M14459; Day 4: number analyzed (Participants) | 33 | 23
  Serogroup B, M14459; Day 4 | 1.99 [1.44 to 2.75] | 1.22 [0.96 to 1.54]
  Serogroup B, M14459; Day 8: number analyzed (Participants) | 33 | 22
  Serogroup B, M14459; Day 8 | 17 [9.31 to 30] | 1.52 [1.05 to 2.20]
  Serogroup B, M14459; Day 31: number analyzed (Participants) | 33 | 45
  Serogroup B, M14459; Day 31 | 24 [14 to 42] | 2.83 [1.88 to 4.24]
  Serogroup B, M01-0240364; Day 1: number analyzed (Participants) | 31 | 44
  Serogroup B, M01-0240364; Day 1 | 2.26 [1.26 to 4.08] | 1.14 [0.97 to 1.35]
  Serogroup B, M01-0240364; Day 4: number analyzed (Participants) | 30 | 23
  Serogroup B, M01-0240364; Day 4 | 2.50 [1.25 to 5.02] | 1.36 [1.02 to 1.82]
  Serogroup B, M01-0240364; Day 8: number analyzed (Participants) | 29 | 21
  Serogroup B, M01-0240364; Day 8 | 525 [257 to 1074] | 1.65 [0.79 to 3.43]
  Serogroup B, M01-0240364; Day 31: number analyzed (Participants) | 30 | 44
  Serogroup B, M01-0240364; Day 31 | 601 [339 to 1064] | 3.05 [1.77 to 5.26]
  Serogroup B, NZ98/254; Day 1 | 1.81 [1.30 to 2.51] | 1.35 [1.15 to 1.59]
  Serogroup B, NZ98/254; Day 4: number analyzed (Participants) | 33 | 23
  Serogroup B, NZ98/254; Day 4 | 1.90 [1.41 to 2.57] | 1.89 [1.38 to 2.59]
  Serogroup B, NZ98/254; Day 8: number analyzed (Participants) | 33 | 22
  Serogroup B, NZ98/254; Day 8 | 8.19 [5.45 to 12] | 1.52 [1.12 to 2.06]
  Serogroup B, NZ98/254; Day 31 | 13 [8.50 to 18] | 3.57 [2.37 to 5.38]
  Serogroup B, M10713; Day 1 | 3.66 [2.38 to 5.62] | 2.56 [1.74 to 3.75]
  Serogroup B, M10713; Day 4: number analyzed (Participants) | 32 | 23
  Serogroup B, M10713; Day 4 | 4.16 [2.70 to 6.41] | 3.73 [2.10 to 6.65]
  Serogroup B, M10713; Day 8: number analyzed (Participants) | 33 | 22
  Serogroup B, M10713; Day 8 | 15 [9.26 to 23] | 2.03 [1.30 to 3.17]
  Serogroup B, M10713; Day 31 | 20 [13 to 31] | 5.51 [3.45 to 8.79]
  Serogroup B, H44/76; Day 1 | 2.33 [1.57 to 3.45] | 1.21 [1.03 to 1.42]
  Serogroup B, H44/76; Day 4: number analyzed (Participants) | 33 | 23
  Serogroup B, H44/76; Day 4 | 2.58 [1.78 to 3.75] | 1.38 [1.05 to 1.81]
  Serogroup B, H44/76; Day 8: number analyzed (Participants) | 33 | 22
  Serogroup B, H44/76; Day 8 | 64 [38 to 109] | 1.84 [1.18 to 2.89]
  Serogroup B, H44/76; Day 31 | 98 [57 to 170] | 5.78 [3.59 to 9.31]
  Serogroup B, 5/99; Day 1 | 13 [7.29 to 22] | 1.78 [1.36 to 2.34]
  Serogroup B, 5/99; Day 4: number analyzed (Participants) | 33 | 23
  Serogroup B, 5/99; Day 4 | 17 [9.56 to 31] | 1.99 [1.36 to 2.92]
  Serogroup B, 5/99; Day 8: number analyzed (Participants) | 33 | 22
  Serogroup B, 5/99; Day 8 | 1768 [1204 to 2596] | 1.97 [0.88 to 4.42]
  Serogroup B, 5/99; Day 31 | 1426 [940 to 2164] | 19 [11 to 34]
  Serogroup A; Day 1 | 4.06 [2.22 to 7.44] | 6.64 [3.56 to 12]
  Serogroup A; Day 4: number analyzed (Participants) | 33 | 23
  Serogroup A; Day 4 | 3.85 [2.00 to 7.42] | 9.69 [3.90 to 24]
  Serogroup A; Day 8: number analyzed (Participants) | 33 | 22
  Serogroup A; Day 8 | 474 [321 to 701] | 61 [25 to 146]
  Serogroup A; Day 31 | 396 [288 to 545] | 149 [106 to 210]
  Serogroup C; Day 1: number analyzed (Participants) | 32 | 46
  Serogroup C; Day 1 | 17 [7.80 to 37] | 6.62 [4.10 to 11]
  Serogroup C; Day 4: number analyzed (Participants) | 30 | 22
  Serogroup C; Day 4 | 21 [9.93 to 43] | 12 [5.13 to 29]
  Serogroup C; Day 8: number analyzed (Participants) | 29 | 19
  Serogroup C; Day 8 | 2664 [1840 to 3855] | 1710 [979 to 2985]
  Serogroup C; Day 31: number analyzed (Participants) | 30 | 38
  Serogroup C; Day 31 | 1676 [1164 to 2414] | 1199 [849 to 1692]
  Serogroup W; Day 1: number analyzed (Participants) | 32 | 46
  Serogroup W; Day 1 | 28 [15 to 53] | 25 [15 to 40]
  Serogroup W; Day 4: number analyzed (Participants) | 25 | 22
  Serogroup W; Day 4 | 19 [8.77 to 41] | 20 [8.11 to 51]
  Serogroup W; Day 8: number analyzed (Participants) | 25 | 16
  Serogroup W; Day 8 | 1285 [900 to 1833] | 1693 [924 to 3103]
  Serogroup W; Day 31: number analyzed (Participants) | 28 | 38
  Serogroup W; Day 31 | 1823 [1163 to 2856] | 2259 [1678 to 3041]
  Serogroup Y; Day 1: number analyzed (Participants) | 32 | 44
  Serogroup Y; Day 1 | 6.17 [3.00 to 13] | 12 [6.29 to 22]
  Serogroup Y; Day 4: number analyzed (Participants) | 31 | 22
  Serogroup Y; Day 4 | 6.53 [3.05 to 14] | 9.60 [3.56 to 26]
  Serogroup Y; Day 8: number analyzed (Participants) | 23 | 13
  Serogroup Y; Day 8 | 722 [429 to 1216] | 1133 [710 to 1809]
  Serogroup Y; Day 31: number analyzed (Participants) | 23 | 23
  Serogroup Y; Day 31 | 779 [430 to 1413] | 1692 [1206 to 2373]

15. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMTs at Day 1, 31, 34, 38, 61 as measure of the kinetics of the immune response following a dose of MenABCWY+OMV, in subjects who were not primed with any meningococcal vaccine (i.e., Naïve Group). This outcome measure reports data for only the Naïve Group as per protocol. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Days 1, 31, 34, 38 and 61
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Naive Group
Number analyzed (Participants) | 50
Titers
  Serogroup B, M14459; Day 1 | 1.48 [1.18 to 1.85]
  Serogroup B, M14459; Day 31 | 4.02 [2.67 to 6.06]
  Serogroup B, M14459; Day 34: number analyzed (Participants) | 26
  Serogroup B, M14459; Day 34 | 5.06 [2.96 to 8.66]
  Serogroup B, M14459; Day 38: number analyzed (Participants) | 24
  Serogroup B, M14459; Day 38 | 9.16 [5.35 to 16]
  Serogroup B, M14459; Day 61: number analyzed (Participants) | 49
  Serogroup B, M14459; Day 61 | 9.78 [6.42 to 15]
  Serogroup B, M01-0240364; Day 1 | 1.23 [1.02 to 1.47]
  Serogroup B, M01-0240364; Day 31: number analyzed (Participants) | 45
  Serogroup B, M01-0240364; Day 31 | 3.11 [1.76 to 5.51]
  Serogroup B, M01-0240364; Day 34: number analyzed (Participants) | 25
  Serogroup B, M01-0240364; Day 34 | 5.13 [2.171 to 12]
  Serogroup B, M01-0240364; Day 38: number analyzed (Participants) | 22
  Serogroup B, M01-0240364; Day 38 | 75 [29 to 199]
  Serogroup B, M01-0240364; Day 61: number analyzed (Participants) | 47
  Serogroup B, M01-0240364; Day 61 | 21 [11 to 38]
  Serogroup B, NZ98/254; Day 1 | 1.45 [1.18 to 1.77]
  Serogroup B, NZ98/254; Day 31 | 5.75 [3.95 to 8.37]
  Serogroup B, NZ98/254; Day 34: number analyzed (Participants) | 26
  Serogroup B, NZ98/254; Day 34 | 6.93 [4.02 to 12]
  Serogroup B, NZ98/254; Day 38: number analyzed (Participants) | 24
  Serogroup B, NZ98/254; Day 38 | 7.92 [5.03 to 12]
  Serogroup B, NZ98/254; Day 61: number analyzed (Participants) | 49
  Serogroup B, NZ98/254; Day 61 | 7.50 [5.12 to 11]
  Serogroup B, M10713; Day 1 | 3.10 [2.16 to 4.45]
  Serogroup B, M10713; Day 31 | 7.70 [5.04 to 12]
  Serogroup B, M10713; Day 34: number analyzed (Participants) | 23
  Serogroup B, M10713; Day 34 | 6.70 [3.37 to 13]
  Serogroup B, M10713; Day 38: number analyzed (Participants) | 24
  Serogroup B, M10713; Day 38 | 8.94 [4.91 to 16]
  Serogroup B, M10713; Day 61: number analyzed (Participants) | 49
  Serogroup B, M10713; Day 61 | 8.73 [5.80 to 13]
  Serogroup B, H44/76; Day 1 | 1.44 [1.14 to 1.80]
  Serogroup B, H44/76; Day 31 | 7.27 [4.53 to 12]
  Serogroup B, H44/76; Day 34: number analyzed (Participants) | 26
  Serogroup B, H44/76; Day 34 | 8.91 [4.62 to 17]
  Serogroup B, H44/76; Day 38: number analyzed (Participants) | 24
  Serogroup B, H44/76; Day 38 | 35 [20 to 60]
  Serogroup B, H44/76; Day 61: number analyzed (Participants) | 49
  Serogroup B, H44/76; Day 61 | 32 [21 to 49]
  Serogroup B, 5/99; Day 1 | 1.90 [1.42 to 2.53]
  Serogroup B, 5/99; Day 31 | 25 [15 to 42]
  Serogroup B, 5/99; Day 34: number analyzed (Participants) | 26
  Serogroup B, 5/99; Day 34 | 40 [18 to 90]
  Serogroup B, 5/99; Day 38: number analyzed (Participants) | 24
  Serogroup B, 5/99; Day 38 | 432 [273 to 683]
  Serogroup B, 5/99; Day 61: number analyzed (Participants) | 49
  Serogroup B, 5/99; Day 61 | 256 [194 to 338]
  Serogroup A; Day 1 | 1.20 [1.05 to 1.37]
  Serogroup A; Day 31 | 22 [14 to 35]
  Serogroup A; Day 34: number analyzed (Participants) | 26
  Serogroup A; Day 34 | 31 [15 to 67]
  Serogroup A; Day 38: number analyzed (Participants) | 24
  Serogroup A; Day 38 | 107 [64 to 179]
  Serogroup A; Day 61: number analyzed (Participants) | 47
  Serogroup A; Day 61 | 74 [51 to 108]
  Serogroup C; Day 1: number analyzed (Participants) | 49
  Serogroup C; Day 1 | 5.11 [3.49 to 7.48]
  Serogroup C; Day 31: number analyzed (Participants) | 48
  Serogroup C; Day 31 | 58 [35 to 96]
  Serogroup C; Day 34: number analyzed (Participants) | 20
  Serogroup C; Day 34 | 94 [54 to 162]
  Serogroup C; Day 38: number analyzed (Participants) | 22
  Serogroup C; Day 38 | 259 [149 to 449]
  Serogroup C; Day 61: number analyzed (Participants) | 47
  Serogroup C; Day 61 | 188 [132 to 266]
  Serogroup W; Day 1: number analyzed (Participants) | 47
  Serogroup W; Day 1 | 8.37 [4.78 to 15]
  Serogroup W; Day 31: number analyzed (Participants) | 46
  Serogroup W; Day 31 | 117 [83 to 166]
  Serogroup W; Day 34: number analyzed (Participants) | 19
  Serogroup W; Day 34 | 180 [107 to 305]
  Serogroup W; Day 38: number analyzed (Participants) | 20
  Serogroup W; Day 38 | 188 [129 to 272]
  Serogroup W; Day 61: number analyzed (Participants) | 41
  Serogroup W; Day 61 | 168 [129 to 218]
  Serogroup Y; Day 1: number analyzed (Participants) | 47
  Serogroup Y; Day 1 | 2.00 [1.40 to 2.85]
  Serogroup Y; Day 31: number analyzed (Participants) | 46
  Serogroup Y; Day 31 | 85 [45 to 163]
  Serogroup Y; Day 34: number analyzed (Participants) | 23
  Serogroup Y; Day 34 | 109 [55 to 215]
  Serogroup Y; Day 38: number analyzed (Participants) | 20
  Serogroup Y; Day 38 | 299 [180 to 495]
  Serogroup Y; Day 61: number analyzed (Participants) | 43
  Serogroup Y; Day 61 | 224 [147 to 343]

16. Secondary Outcome: GMR Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMRs as measure of the kinetics of the immune response following a dose of MenABCWY+OMV, in subjects who previously received 2 doses of MenABCWY+OMV or 1 dose of MenACWY. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Days 4, 8 and 31 versus Day 1.
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | MenABCWY+OMV Group | MenACWY Group
Number analyzed (Participants) | 33 | 46
Ratios
  Serogroup B, M14459; Dy 4/Day 1: number analyzed (Participants) | 33 | 23
  Serogroup B, M14459; Dy 4/Day 1 | 0.98 [0.88 to 1.09] | 0.80 [0.60 to 1.05]
  Serogroup B, M14459; Day 8/Day 1: number analyzed (Participants) | 33 | 22
  Serogroup B, M14459; Day 8/Day 1 | 8.19 [4.58 to 15] | 1.21 [0.80 to 1.83]
  Serogroup B, M14459; Day 31/Day 1: number analyzed (Participants) | 33 | 45
  Serogroup B, M14459; Day 31/Day 1 | 12 [6.88 to 20] | 2.11 [1.45 to 3.07]
  Serogroup B, M01-0240364; Day 4/Day 1: number analyzed (Participants) | 30 | 22
  Serogroup B, M01-0240364; Day 4/Day 1 | 1.08 [0.68 to 1.71] | 1.06 [0.90 to 1.25]
  Serogroup B, M01-0240364; Day 8/Day 1: number analyzed (Participants) | 28 | 20
  Serogroup B, M01-0240364; Day 8/Day 1 | 210 [85 to 517] | 1.69 [0.78 to 3.66]
  Serogroup B, M01-0240364; Day 31/Day 1: number analyzed (Participants) | 28 | 42
  Serogroup B, M01-0240364; Day 31/Day 1 | 229 [108 to 485] | 2.80 [1.59 to 4.96]
  Serogroup B, NZ98/254; Day 4/Day 1: number analyzed (Participants) | 33 | 23
  Serogroup B, NZ98/254; Day 4/Day 1 | 1.05 [0.84 to 1.31] | 1.19 [0.90 to 1.58]
  Serogroup B, NZ98/254; Day 8/Day 1: number analyzed (Participants) | 33 | 22
  Serogroup B, NZ98/254; Day 8/Day 1 | 4.53 [2.93 to 7.02] | 1.31 [0.90 to 1.90]
  Serogroup B, NZ98/254; Day 31/Day 1 | 6.92 [4.61 to 10] | 2.64 [1.73 to 4.02]
  Serogroup B, M10713; Day 4/Day 1: number analyzed (Participants) | 32 | 23
  Serogroup B, M10713; Day 4/Day 1 | 1.09 [0.93 to 1.28] | 0.93 [0.76 to 1.14]
  Serogroup B, M10713; Day 8/Day 1: number analyzed (Participants) | 33 | 22
  Serogroup B, M10713; Day 8/Day 1 | 4.02 [2.74 to 5.88] | 1.22 [0.89 to 1.67]
  Serogroup B, M10713; Day 31/Day 1 | 5.38 [3.54 to 8.17] | 2.15 [1.46 to 3.17]
  Serogroup B, H44/76; Day 4/Day 1: number analyzed (Participants) | 33 | 23
  Serogroup B, H44/76; Day 4/Day 1 | 1.11 [0.88 to 1.4128] | 1.00 [0.79 to 1.27]
  Serogroup B, H44/76; Day 8/Day 1: number analyzed (Participants) | 33 | 22
  Serogroup B, H44/76; Day 8/Day 1 | 28 [15 to 50] | 1.73 [1.06 to 2.81]
  Serogroup B, H44/76; Day 31/Day 1 | 42 [25 to 72] | 4.78 [2.90 to 7.89]
  Serogroup B, 5/99; Day 4/Day 1: number analyzed (Participants) | 33 | 23
  Serogroup B, 5/99; Day 4/Day 1 | 1.35 [0.90 to 2.04] | 0.93 [0.68 to 1.26]
  Serogroup B, 5/99; Day 8/Day 1: number analyzed (Participants) | 33 | 22
  Serogroup B, 5/99; Day 8/Day 1 | 139 [77 to 248] | 1.30 [0.66 to 2.57]
  Serogroup B, 5/99; Day 31/Day 1 | 112 [68 to 185] | 11 [6.09 to 19]
  Serogroup A; Day 4/Day 1: number analyzed (Participants) | 33 | 23
  Serogroup A; Day 4/Day 1 | 0.95 [0.72 to 1.24] | 0.87 [0.61 to 1.24]
  Serogroup A; Day 8/Day 1: number analyzed (Participants) | 33 | 22
  Serogroup A; Day 8/Day 1 | 117 [59 to 232] | 17 [7.78 to 37]
  Serogroup A; Day 31/Day 1 | 98 [54 to 177] | 22 [13 to 38]
  Serogroup C; Day 4/Day 1: number analyzed (Participants) | 29 | 22
  Serogroup C; Day 4/Day 1 | 1.30 [0.98 to 1.73] | 1.20 [0.92 to 1.56]
  Serogroup C; Day 8/Day 1: number analyzed (Participants) | 28 | 19
  Serogroup C; Day 8/Day 1 | 164 [65 to 411] | 491 [211 to 1141]
  Serogroup C; Day 31/Day 1: number analyzed (Participants) | 30 | 38
  Serogroup C; Day 31/Day 1 | 105 [49 to 222] | 238 [145 to 392]
  Serogroup W; Day 4/Day 1: number analyzed (Participants) | 25 | 22
  Serogroup W; Day 4/Day 1 | 0.90 [0.56 to 1.442] | 0.97 [0.68 to 1.37]
  Serogroup W; Day 8/Day 1: number analyzed (Participants) | 24 | 16
  Serogroup W; Day 8/Day 1 | 61 [29 to 131] | 67 [27 to 168]
  Serogroup W; Day 31/Day 1: number analyzed (Participants) | 28 | 38
  Serogroup W; Day 31/Day 1 | 67 [34 to 132] | 112 [65 to 191]
  Serogroup Y; Day 4/Day 1: number analyzed (Participants) | 30 | 22
  Serogroup Y; Day 4/Day 1 | 1.06 [0.79 to 1.41] | 0.73 [0.49 to 1.09]
  Serogroup Y; Day 8/Day 1: number analyzed (Participants) | 22 | 13
  Serogroup Y; Day 8/Day 1 | 156 [62 to 390] | 132 [33 to 535]
  Serogroup Y; Day 31/Day 1: number analyzed (Participants) | 22 | 22
  Serogroup Y; Day 31/Day 1 | 162 [70 to 375] | 216 [80 to 580]

17. Secondary Outcome: GMR Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMRs as measure of the kinetics of the immune response following a dose of MenABCWY+OMV, in Naïve subjects. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Days 31, 34, 38 and 61 versus Day 1.
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | Naive Group
Number analyzed (Participants) | 50
Ratios
  Serogroup B, M14459; Day 31/Day 1 | 2.72 [1.91 to 3.87]
  Serogroup B, M14459; Day 34/Day 1: number analyzed (Participants) | 26
  Serogroup B, M14459; Day 34/Day 1 | 3.45 [2.09 to 5.72]
  Serogroup B, M14459; Day 38/Day 1: number analyzed (Participants) | 24
  Serogroup B, M14459; Day 38/Day 1 | 6.15 [3.65 to 10]
  Serogroup B, M14459; Day 61/Day 1: number analyzed (Participants) | 49
  Serogroup B, M14459; Day 61/Day 1 | 6.78 [4.51 to 10]
  Serogroup B, M01-0240364; Day 31/Day 1: number analyzed (Participants) | 45
  Serogroup B, M01-0240364; Day 31/Day 1 | 2.48 [1.51 to 4.07]
  Serogroup B, M01-0240364; Day 34/Day 1: number analyzed (Participants) | 25
  Serogroup B, M01-0240364; Day 34/Day 1 | 3.97 [1.79 to 8.80]
  Serogroup B, M01-0240364; Day 38/Day 1: number analyzed (Participants) | 22
  Serogroup B, M01-0240364; Day 38/Day 1 | 64 [24 to 167]
  Serogroup B, M01-0240364; Day 61/Day 1: number analyzed (Participants) | 47
  Serogroup B, M01-0240364; Day 61/Day 1 | 18 [9.90 to 33]
  Serogroup B, NZ98/254; Day 31/Day 1 | 3.98 [2.73 to 5.79]
  Serogroup B, NZ98/254; Day 34/Day 1: number analyzed (Participants) | 26
  Serogroup B, NZ98/254; Day 34/Day 1 | 4.52 [2.60 to 7.84]
  Serogroup B, NZ98/254; Day 38/Day 1: number analyzed (Participants) | 24
  Serogroup B, NZ98/254; Day 38/Day 1 | 5.84 [3.34 to 10]
  Serogroup B, NZ98/254; Day 61/Day 1: number analyzed (Participants) | 49
  Serogroup B, NZ98/254; Day 61/Day 1 | 5.28 [3.61 to 7.74]
  Serogroup B, M10713; Day 31/Day 1 | 2.48 [1.78 to 3.45]
  Serogroup B, M10713; Day 34/Day 1: number analyzed (Participants) | 23
  Serogroup B, M10713; Day 34/Day 1 | 2.54 [1.67 to 3.86]
  Serogroup B, M10713; Day 38/Day 1: number analyzed (Participants) | 24
  Serogroup B, M10713; Day 38/Day 1 | 2.83 [1.64 to 4.87]
  Serogroup B, M10713; Day 61/Day 1: number analyzed (Participants) | 49
  Serogroup B, M10713; Day 61/Day 1 | 2.85 [1.98 to 4.11]
  Serogroup B, H44/76; Day 31/Day 1 | 5.06 [3.21 to 7.97]
  Serogroup B, H44/76; Day 34/Day 1: number analyzed (Participants) | 26
  Serogroup B, H44/76; Day 34/Day 1 | 6.17 [3.33 to 11]
  Serogroup B, H44/76; Day 38/Day 1: number analyzed (Participants) | 24
  Serogroup B, H44/76; Day 38/Day 1 | 24 [14 to 42]
  Serogroup B, H44/76; Day 61/Day 1: number analyzed (Participants) | 49
  Serogroup B, H44/76; Day 61/Day 1 | 23 [15 to 35]
  Serogroup B, 5/99; Day 31/Day 1 | 13 [8.14 to 22]
  Serogroup B, 5/99; Day 34/Day 1: number analyzed (Participants) | 26
  Serogroup B, 5/99; Day 34/Day 1 | 20 [8.58 to 49]
  Serogroup B, 5/99; Day 38/Day 1: number analyzed (Participants) | 24
  Serogroup B, 5/99; Day 38/Day 1 | 233 [141 to 385]
  Serogroup B, 5/99; Day 61/Day 1: number analyzed (Participants) | 49
  Serogroup B, 5/99; Day 61/Day 1 | 141 [106 to 189]
  Serogroup A; Day 31/Day 1 | 18 [12 to 29]
  Serogroup A; Day 34/Day 1: number analyzed (Participants) | 26
  Serogroup A; Day 34/Day 1 | 28 [13 to 61]
  Serogroup A; Day 38/Day 1: number analyzed (Participants) | 24
  Serogroup A; Day 38/Day 1 | 82 [48 to 140]
  Serogroup A; Day 61/Day 1: number analyzed (Participants) | 47
  Serogroup A; Day 61/Day 1 | 61 [41 to 90]
  Serogroup C; Day 31/Day 1: number analyzed (Participants) | 48
  Serogroup C; Day 31/Day 1 | 12 [6.88 to 19]
  Serogroup C; Day 34/Day 1: number analyzed (Participants) | 19
  Serogroup C; Day 34/Day 1 | 18 [8.98 to 36]
  Serogroup C; Day 38/Day 1: number analyzed (Participants) | 22
  Serogroup C; Day 38/Day 1 | 64 [32 to 128]
  Serogroup C; Day 61/Day 1: number analyzed (Participants) | 46
  Serogroup C; Day 61/Day 1 | 39 [25 to 61]
  Serogroup W; Day 31/Day 1: number analyzed (Participants) | 44
  Serogroup W; Day 31/Day 1 | 16 [8.35 to 30]
  Serogroup W; Day 34/Day 1: number analyzed (Participants) | 18
  Serogroup W; Day 34/Day 1 | 42 [15 to 116]
  Serogroup W; Day 38/Day 1: number analyzed (Participants) | 19
  Serogroup W; Day 38/Day 1 | 16 [6.68 to 40]
  Serogroup W; Day 61/Day 1: number analyzed (Participants) | 38
  Serogroup W; Day 61/Day 1 | 22 [11 to 42]
  Serogroup Y; Day 31/Day 1: number analyzed (Participants) | 43
  Serogroup Y; Day 31/Day 1 | 46 [23 to 92]
  Serogroup Y; Day 34/Day 1: number analyzed (Participants) | 20
  Serogroup Y; Day 34/Day 1 | 69 [30 to 1601]
  Serogroup Y; Day 38/Day 1: number analyzed (Participants) | 20
  Serogroup Y; Day 38/Day 1 | 134 [68 to 264]
  Serogroup Y; Day 61/Day 1: number analyzed (Participants) | 40
  Serogroup Y; Day 61/Day 1 | 106 [62 to 182]

18. Secondary Outcome: Percentages of Subjects With hSBA ≥ LLQ Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: The HT-hSBA assay format was changed in 2015 in response to CBER comments and no new LLQ values were defined as the validation of this format was not relevant. The LLQ cut off values for the old assay format correspond to 8 for serogroups A,C,W and Y and 5 for serogroup B strains and these results are presented in outcome measures 19 and 20 and are considered final in Company's judgement.
Time Frame: At Day 61
Population: Data was not collected for this outcome measure as validation procedure of the hSBA assay was not relevant to the study.
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Percentages of Subjects With hSBA ≥ 8 Against N. Meningitidis Serogroups A, C, W and Y.
Description: Immunogenicity against N. meningitidis serogroup A, C, W and Y following 2 doses of MenABCWY+OMV in subjects who previously received 1 dose of MenACWY and Naïve subjects, at Day 61, as measured by percentages of subjects with hSBA ≥ 8.
Time Frame: At Day 61
Population: Analysis was performed on Full Analysis Set immunogenicity persistence population set Day 61- all subjects in the enrolled population who received a study vaccination, provided at least one evaluable serum sample at 1 month post second vaccination and whose assay result was available for at least one serogroup/ test strain
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 46 | 47
Percentages of subjects
  Serogroup A | 100 [92.3 to 100.0] | 94 [82.5 to 98.7]
  Serogroup C: number analyzed (Participants) | 34 | 47
  Serogroup C | 100 [89.7 to 100.0] | 100 [92.5 to 100.0]
  Serogroup W: number analyzed (Participants) | 32 | 41
  Serogroup W | 100 [89.1 to 100.0] | 100 [91.4 to 100.0]
  Serogroup Y: number analyzed (Participants) | 27 | 43
  Serogroup Y | 100 [87.2 to 100.0] | 98 [87.7 to 99.94]

20. Secondary Outcome: Percentages of Subjects With hSBA ≥ 5 Against N. Meningitidis Serogroup B Test Strains.
Description: Immunogenicity against N. meningitidis serogroup B test strains following 2 doses of MenABCWY+OMV in subjects who previously received 1 dose of MenACWY and Naïve subjects, at Day 61, as measured by percentages of subjects with hSBA ≥ 5. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Day 61
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 46 | 49
Percentages of subjects
  Serogroup B, M14459 | 46 [30.9 to 61.0] | 67 [52.5 to 80.1]
  Serogroup B, M01-0240364: number analyzed (Participants) | 46 | 47
  Serogroup B, M01-0240364 | 65 [49.8 to 78.6] | 70 [55.1 to 82.7]
  Serogroup B, NZ98/254 | 46 [30.9 to 61.0] | 61 [46.2 to 74.8]
  Serogroup B, M10713 | 54 [39.0 to 69.1] | 65 [50.4 to 78.3]
  Serogroup B, H44/76 | 85 [71.1 to 93.7] | 88 [75.2 to 95.4]
  Serogroup B, 5/99 | 100 [92.3 to 100.0] | 100 [92.7 to 100.0]

21. Secondary Outcome: GMTs Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMTs as measure of the immunogenicity of 2 doses of MenABCWY+OMV in subjects who previously received 1 dose of MenACWY and Naïve subjects, at Day 61. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: At Day 61
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 46 | 49
Titers
  Serogroup B, M14459 | 4.82 [3.26 to 7.12] | 9.78 [6.42 to 15]
  Serogroup B, M01-0240364: number analyzed (Participants) | 46 | 47
  Serogroup B, M01-0240364 | 19 [10 to 34] | 21 [11 to 38]
  Serogroup B, NZ98/254 | 6.24 [4.47 to 8.70] | 7.50 [5.12 to 11]
  Serogroup B, M10713 | 6.91 [4.43 to 11] | 8.73 [5.80 to 13]
  Serogroup B, H44/76 | 19 [13 to 28] | 32 [21 to 49]
  Serogroup B, 5/99 | 196 [149 to 257] | 256 [194 to 338]
  Serogroup A: number analyzed (Participants) | 46 | 47
  Serogroup A | 222 [170 to 290] | 74 [51 to 108]
  Serogroup C: number analyzed (Participants) | 34 | 47
  Serogroup C | 879 [712 to 1085] | 188 [132 to 266]
  Serogroup W: number analyzed (Participants) | 32 | 41
  Serogroup W | 1440 [1078 to 1924] | 168 [129 to 218]
  Serogroup Y: number analyzed (Participants) | 27 | 43
  Serogroup Y | 1576 [1190 to 2087] | 224 [147 to 343]
Statistical Analysis 1: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis Serogroup B, M14459; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.49, 95% CI 2-sided [0.28 to 0.87]
Statistical Analysis 2: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis Serogroup B, M01-0240364; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.91, 95% CI 2-sided [0.40 to 2.11]
Statistical Analysis 3: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup B, NZ98/254; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.83, 95% CI 2-sided [0.50 to 1.38]
Statistical Analysis 4: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup B, M10713; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.79, 95% CI 2-sided [0.44 to 1.44]
Statistical Analysis 5: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup B, H44/76; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.60, 95% CI 2-sided [0.34 to 1.07]
Statistical Analysis 6: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup B, 5/99; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 0.77, 95% CI 2-sided [0.52 to 1.12]
Statistical Analysis 7: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup A; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 2.99, 95% CI 2-sided [1.89 to 4.75]
Statistical Analysis 8: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup C; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 4.69, 95% CI 2-sided [3.01 to 7.31]
Statistical Analysis 9: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup W; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 8.60, 95% CI 2-sided [5.84 to 13]
Statistical Analysis 10: Comparison: MenACWY Group vs Naive Group; Between-group GMT ratios against N. meningitidis serogroup Y; Test type: Other; Miettinen & Nurminen score method; Geometric mean ratio = 7.03, 95% CI 2-sided [3.96 to 12]

22. Secondary Outcome: GMRs Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains.
Description: GMRs as measure of the immunogenicity of 2 doses of MenABCWY+OMV in subjects who previously received 1 dose of MenACWY and Naïve subjects. The Meningococcal B Strains were M14459, M01-0240364, NZ98/254, M10713, H44/76 and 5/99.
Time Frame: Day 61 versus Day 1 (baseline)
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 46 | 49
Ratios
  Serogroup B, M14459 | 3.50 [2.33 to 5.26] | 6.78 [4.51 to 10]
  Serogroup B, M01-0240364: number analyzed (Participants) | 44 | 47
  Serogroup B, M01-0240364 | 16 [8.77 to 31] | 18 [9.90 to 33]
  Serogroup B, NZ98/254 | 4.61 [3.22 to 6.60] | 5.28 [3.61 to 7.74]
  Serogroup B, M10713 | 2.70 [1.94 to 3.77] | 2.85 [1.98 to 4.11]
  Serogroup B, H44/76 | 16 [10 to 24] | 23 [15 to 35]
  Serogroup B, 5/99 | 110 [76 to 159] | 141 [106 to 189]
  Serogroup A: number analyzed (Participants) | 46 | 47
  Serogroup A | 33 [20 to 56] | 61 [41 to 90]
  Serogroup C: number analyzed (Participants) | 34 | 46
  Serogroup C | 181 [108 to 303] | 39 [25 to 61]
  Serogroup W: number analyzed (Participants) | 32 | 38
  Serogroup W | 85 [46 to 155] | 22 [11 to 42]
  Serogroup Y: number analyzed (Participants) | 26 | 40
  Serogroup Y | 264 [117 to 598] | 106 [62 to 182]

23. Secondary Outcome: Number of Subjects Reporting Any Unsolicited and Solicited Adverse Events (AEs) Within 30 Min After Each Vaccination
Description: Any solicited and unsolicited AEs reported within 30 minutes after each vaccination. Assessed solicited local symptoms were: Erythema and Induration. Any = occurrence of the symptom spreading beyond 25 millimeters (mm) of injection site. Assessed solicited general symptoms were: Arthralgia, Chills, Fatigue, Headache, Loss of Appetite, Myalgia, Nausea and Fever (body temperature ≥ 38°C). Other solicited data included: Prevention of Pain and/or Fever and Treatment of Pain and/or Fever. Any = occurrence of the symptom regardless of intensity grade. Note: There were no unsolicited AEs reported within 30 minutes after vaccination.
Time Frame: Within 30 min after each vaccination
Population: Analysis was performed on Solicited safety Set- included all subjects in the Full Analysis Set Immunogenicity population who provided post-vaccination safety data.
Measure: Number; unit: Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Subjects
  Erythema (1st vaccination) | 0 | 1 | 0
  Erythema (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Erythema (2nd vaccination) |  | 1 | 0
  Induration (1st vaccination) | 0 | 0 | 0
  Induration (2nd vaccination): number analyzed (Participants) | 0 | 46 | 50
  Induration (2nd vaccination) |  | 0 | 0
  Pain (1st vaccination) | 4 | 8 | 6
  Pain (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Pain (2nd vaccination) |  | 3 | 4
  Arthralgia (1st vaccination) | 0 | 0 | 0
  Arthralgia (2nd vaccination): number analyzed (Participants) | 0 | 46 | 50
  Arthralgia (2nd vaccination) |  | 0 | 0
  Chills (1st vaccination) | 0 | 0 | 0
  Chills (2nd vaccination): number analyzed (Participants) | 0 | 46 | 50
  Chills (2nd vaccination) |  | 0 | 0
  Fatigue (1st vaccination) | 0 | 0 | 0
  Fatigue (2nd vaccination): number analyzed (Participants) | 0 | 46 | 50
  Fatigue (2nd vaccination) |  | 0 | 1
  Headache (1st vaccination) | 1 | 0 | 0
  Headache (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Headache (2nd vaccination) |  | 0 | 1
  Loss of Appetite (1st vaccination) | 0 | 0 | 0
  Loss of Appetite (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Loss of Appetite (2nd vaccination) |  | 0 | 0
  Myalgia (1st vaccination) | 0 | 0 | 0
  Myalgia (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Myalgia (2nd vaccination) |  | 0 | 0
  Nausea (1st vaccination) | 0 | 0 | 0
  Nausea (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Nausea (2nd vaccination) |  | 0 | 0
  Fever (1st vaccination) | 0 | 0 | 0
  Fever (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Fever (2nd vaccination) |  | 0 | 0
  Prevention of Pain/Fever (1st vaccination): number analyzed (Participants) | 33 | 45 | 50
  Prevention of Pain/Fever (1st vaccination) | 0 | 0 | 0
  Prevention of Pain/Fever (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Prevention of Pain/Fever (2nd vaccination) |  | 0 | 1
  Treatment of Pain/Fever (1st vaccination): number analyzed (Participants) | 33 | 45 | 50
  Treatment of Pain/Fever (1st vaccination) | 0 | 0 | 0
  Treatment of Pain/Fever (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Treatment of Pain/Fever (2nd vaccination) |  | 0 | 2

24. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were Erythema, Induration and Pain. Any = occurrence of the symptom spreading beyond 25 millimeters (mm) of injection site.
Time Frame: From Day 1 (6 hours) to Day 7 after each vaccination
Population: as for outcome 23
Measure: Number; unit: Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Subjects
  Any local AEs (1st vaccination) | 31 | 41 | 47
  Erythema (1st vaccination): number analyzed (Participants) | 33 | 45 | 50
  Erythema (1st vaccination) | 8 | 7 | 8
  Induration (1st vaccination) | 12 | 7 | 13
  Pain (1st vaccination) | 31 | 41 | 47
  Any local AEs (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Any local AEs (2nd vaccination) |  | 35 | 41
  Erythema (2nd vaccination): number analyzed (Participants) | 0 | 45 | 49
  Erythema (2nd vaccination) |  | 6 | 7
  Induration (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Induration (2nd vaccination) |  | 9 | 8
  Pain (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Pain (2nd vaccination) |  | 34 | 41

25. Secondary Outcome: Number of Subjects With Solicited Systemic Symptoms and Other Solicited Data
Description: Assessed solicited systemic symptoms were Arthralgia, Chills, Fatigue, Headache, Loss of Appetite, Myalgia, Nausea and Fever (body temperature ≥ 38°C). Other solicited data included: Prevention of pain and/or fever and Treatment of pain and/or fever. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: From Day 1 (6 hours) to Day 7 after each vaccination
Population: as for outcome 23
Measure: Number; unit: Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Subjects
  Any systemic AEs (1st vaccination) | 24 | 35 | 37
  Arthralgia (1st vaccination) | 8 | 8 | 15
  Chills (1st vaccination) | 5 | 11 | 11
  Fatigue (1st vaccination): number analyzed (Participants) | 33 | 45 | 50
  Fatigue (1st vaccination) | 14 | 19 | 24
  Headache (1st vaccination) | 19 | 20 | 23
  Loss of Appetite (1st vaccination): number analyzed (Participants) | 33 | 45 | 50
  Loss of Appetite (1st vaccination) | 5 | 9 | 9
  Myalgia (1st vaccination) | 18 | 22 | 23
  Nausea (1st vaccination) | 4 | 10 | 13
  Fever (1st vaccination) | 0 | 4 | 8
  Prevention of Pain/Fever (1st vaccination): number analyzed (Participants) | 33 | 44 | 50
  Prevention of Pain/Fever (1st vaccination) | 0 | 1 | 1
  Treatment of Pain/Fever (1st vaccination): number analyzed (Participants) | 33 | 44 | 50
  Treatment of Pain/Fever (1st vaccination) | 8 | 7 | 11
  Any systemic AEs (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Any systemic AEs (2nd vaccination) |  | 22 | 28
  Arthralgia (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Arthralgia (2nd vaccination) |  | 4 | 7
  Chills (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Chills (2nd vaccination) |  | 5 | 9
  Fatigue (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Fatigue (2nd vaccination) |  | 10 | 12
  Headache (2nd vaccination): number analyzed (Participants) | 0 | 44 | 50
  Headache (2nd vaccination) |  | 11 | 18
  Loss of Appetite (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Loss of Appetite (2nd vaccination) |  | 3 | 5
  Myalgia (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Myalgia (2nd vaccination) |  | 12 | 14
  Nausea (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Nausea (2nd vaccination) |  | 4 | 4
  Fever (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Fever (2nd vaccination) |  | 4 | 2
  Prevention of Pain/Fever (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Prevention of Pain/Fever (2nd vaccination) |  | 1 | 3
  Treatment of Pain/Fever (2nd vaccination): number analyzed (Participants) | 0 | 45 | 50
  Treatment of Pain/Fever (2nd vaccination) |  | 2 | 6

26. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Possibly or Probably related = AE assessed by the investigator as related to the vaccination.
Time Frame: From Day 1 to Day 31 after each vaccination (Day 1 to Day 31 for MenABCWY+OMV Group and Day 1 to Day 61 for MenACWY and Naive Groups)
Population: Analysis was performed on Unsolicited Safety Set- included all subjects in the Exposed Set who had post-vaccination unsolicited adverse event records.
Measure: Number; unit: Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Subjects
  Any AEs | 11 | 21 | 20
  Possibly or Probably Related AEs | 3 | 11 | 8

27. Secondary Outcome: Number of Subjects With Medically Attended AEs Reported During the Entire Study Period.
Description: Medically attended AEs = were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any medically attended AE(s) = Occurrence of any medically attended AE(s) regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (Day 1 to Day 31 for MenABCWY+OMV Group and Day 1 to Day 61 for MenACWY and Naive Groups)
Population: as for outcome 26
Measure: Number; unit: Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Subjects | 2 | 6 | 5

28. Secondary Outcome: Number of Subjects With Unsolicited AEs Leading to Premature Withdrawal From Study Reported During the Entire Study Period.
Description: The number of subjects who reported unsolicited AEs leading to premature withdrawal from study after any vaccination.
Time Frame: From Day 1 to Day 31 (MenABCWY+OMV Group) and from Day 1 to Day 61 (MenACWY and Naive Groups)
Population: as for outcome 26
Measure: Number; unit: Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Subjects | 0 | 1 | 0

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Reported During the Entire Study Period.
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Any SAE(s) = Occurrence of any SAE(s) regardless of intensity grade or relation to vaccination. Possibly or probably related SAE(s) = SAE(s) assessed by the investigator as related to the vaccination.
Time Frame: as for outcome 27
Population: as for outcome 26
Measure: Number; unit: Subjects
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
Number analyzed (Participants) | 33 | 46 | 50
Subjects
  Any SAEs | 0 | 0 | 0
  Possibly or probably related SAEs | 0 | 0 | 0
  AEs leading to death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and systemic symptoms: from Day 1 (6 hours) to Day 7 after each study vaccination; Unsolicited AEs: from Day 1 to Day 31 after each study vaccination; SAEs: during the entire study period (from Day 1 to Day 61).
Arm/Group | MenABCWY+OMV Group | MenACWY Group | Naive Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/46 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/46 | 0/50
Other Adverse Events (participants affected / at risk) | 33/33 | 44/46 | 48/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenABCWY+OMV Group (N=33) | MenACWY Group (N=46) | Naive Group (N=50)
Headache (Nervous system disorders) | 19 (43) | 23 (84) | 28 (120)
Chills (General disorders) | 5 (10) | 14 (25) | 16 (31)
Fatigue (General disorders) | 14 (29) | 20 (75) | 27 (82)
Injection site erythema (General disorders) | 11 (45) | 26 (135) | 30 (123)
Injection site induration (General disorders) | 18 (75) | 27 (173) | 30 (169)
Injection site pain (General disorders) | 31 (114) | 42 (295) | 48 (333)
Pyrexia (General disorders) | 0 (0) | 8 (12) | 10 (13)
Nausea (Gastrointestinal disorders) | 4 (11) | 10 (30) | 15 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14) | 11 (35) | 19 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (42) | 25 (85) | 26 (96)
Decreased appetite (Metabolism and nutrition disorders) | 5 (11) | 11 (25) | 13 (30)
Nasopharyngitis (Infections and infestations) | 1 (1) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.